CLINICAL TRIAL: NCT06649032
Title: A Multicentric Epidemiological Study of the Actual Incidence of Respiratory Tract Infections in an Adult Italian Population, With or Without Underlying Risk Factors
Brief Title: Survey of Incidence of Respiratory Tract Infections
Acronym: SIRTI
Status: Completed | Type: Observational
Sponsor: Lallemand Pharma AG (Industry)
Collaborators: Istituto di Farmacologia Traslazionale - National Research Council (IFT-CNR) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023/09/01
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Healthy Adults; Not Healthy Adults
Keywords: incidence; adults; respiratory tract infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort Incidence: This cohort will comprise subjects recruited from 1st November 2023 to 21st December 2023 and followed from 22nd December 2023 to 30th April 2024 and subjects recruited from 01st November 2024 to 21st December 2024 and followed from 22nd Dec 2024 to 30th April 2025. During the follow-up period, the subjects will be asked to report respiratory tract infections to the investigators (phone calls or study visit).
  Interventions: Other: No intervention
- Cohort Respiratory Tract Infections (RTI) positive: Subjects recruited from 1st November 2023 to 21st December 2023, followed from 22nd December 2023 to 30th April 2024 and who developed at least one respiratory tract infection will be also followed from 22nd December 2024 to 30th April 2025 and asked to report respiratory tract infections to the investigators.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no difference: both cohorts are followed in the same way

SUMMARY:
The purpose of this study is to acquire reliable and current data on the actual incidence (post-COVID) of respiratory tract infections in the general adult population in the absence of any intervention. These data will provide useful background information for designing future studies aimed at assessing whether preventive measures or pharmacological treatments are beneficial in reducing the frequency and severity of infectious episodes.

DETAILED DESCRIPTION:
This multicentric prospective observational survey will be carried out in Italy during the winter and early spring ( December 22nd to April 30th) in two consecutive years on approximately 2750 subjects recruited in the period between November 1st and December 21st in different medical settings and regions.

Investigators from 4 different institutions will be involved:

FIMMG (Federazione Italiana dei Medici di Medicina Generale). Ten general practitioners will recruit approx. 1000 consecutive subjects from the general population.

SIAAIC (Societa' Italiana di Allergologia, Asma e Immunologia Clkinica). Ten allergy specialists will recruit approx.1000 consecutive subjects suffering from allergic diseases.

Fondazione Maugeri (5 Centers) and UCSC (Universita' Cattolica del Sacro Cuore) / Policlinico Gemelli will recruit approx. 750 consecutive subjects suffering from asthma or COPD.

Participants having signed an informed consent at any suspected Respiratory Tract Infection (RTI) during the observation period will be asked to contact (phone call or visit) the investigator to record the relevant clinical information documenting the RTI episode.

At the end of the observation period all subjects will be contacted by the investigators to check for completeness and compliance of the RTI reporting.

The procedure will be repeated in the same way in the second year of survey but including subjects having experienced at least one confirmed RTI during the first year. This will allow assessing intra-individual variability of infectious episodes from year to year.

ELIGIBILITY:
Inclusion Criteria:

Male or female aged from at least 18 years -

Exclusion Criteria:

Minor subjects-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: During both enrolment periods, the study participation will be proposed to adults (without risk factors for respiratory tract infections or with risk factor, e.g. asthma, allergy, COPD) visiting their practitioner for any medical reason. During the observation periods, the subjects who accept study participation will report respiratory tract infections to the investigators.
Sampling Method: Non-Probability Sample
Enrollment: 1736 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Incidence of respiratory tract infections during the whole observation period (whole population, with risk factor, without risk factor) | From 22nd Dec 2023 to 30th Apr2024 and from 22nd Dec 2024 to 30th Apr 2025
  Overall mean number of respiratory tract infections during both observation periods (whole period), mean number of respiratory tract infections for subjects with or without risk factors during the whole period.

SECONDARY OUTCOMES:
Number of subjects of the Cohort Incidence with at least one respiratory tract infection during the first observation period (whole population, with risk factor, without risk factor) | from 22nd Dec 2023 to 30th Apr 2024
Number of subjects of the Cohort Incidence with at least one respiratory tract infection during the second observation period (whole population, with risk factor, without risk factor) | from 22nd Dec 2024 to 30th Apr 2025
Number of subjects from the Cohort RTI positive who had at least one respiratory tract infection during the second observation period | From 22nd Dec 2024 to 30th Apr 2025
Total and mean number of respiratory tract infections during the first observation period for subjects belonging to the Cohort Incidence (whole population, with risk factor, without risk factor) | from 22nd Dec 2023 to 30th Apr 2024
Total and mean number of respiratory tract infections during the second observation period for subjects belonging to the Cohort Incidence (whole population, with risk factor, without risk factor) | from 22nd Dec 2024 to 30th Apr 2025
Comparaison of the mean number of respiratory tract infections during the first observation period versus the second one for subjects belonging to the Cohort RTI positive (whole population, with risk factor, without risk factor) | from 22nd Dec 2023 to 30th Apr 2024 and from 22nd Dec 2024 to 30th Apr 2025
Total and mean number of respiratory tract infections during the first observation period for subjects belonging to the Cohort RTI positive (whole population, with risk factor, without risk factor | from 22nd Dec 2023 to 30th Apr 2024
Total and mean number of respiratory tract infections during the second observation period for subjects belonging to the Cohort RTI positive (whole population, with risk factor, without risk factor) | from 22nd Dec 2024 to 30th Apr 2025
Total and mean number of respiratory tract infections during the whole observation period for subjects belonging to the Cohort RTI positive (whole population, with risk factor, without risk factor) | from 22nd Dec 2023 to 30th Apr 2024 and from 22nd Dec 2024 to 30th Apr 2025
Time to first respiratory infection during the first observation period (whole population, with risk factor, without risk factor) for subjects of the Cohort Incidence | from 22nd Dec 2023 to 30th Apr 2024
Time to first respiratory infection of the subjects belonging to the Cohort Incidence during the second observation period (whole population, with risk factor, without risk factor | from 22nd Dec 2024 to 30th Apr 2025
Time to first respiratory tract infection in the subjects belonging to the Cohort Incidence during the whole observation period (whole population, with risk factor, without risk factor | 023 to 30th Apr 2024 and from 22nd Dec 2024 to 30th Apr 2025 from 22nd Dec 2
Comparaison of the mean number of respiratory tract infections during the first observation period versus the second one for subjects belonging to the Cohort Incidence (whole population, with risk factor, without risk factor) | from 22nd Dec 2023 to 30th Apr 2024 and from 22nd Dec 2024 to 30th Apr 2025
Number of subjects of the Cohort RTI positive with recurrent respiratory tract infections (≥2) during each consecutive observation period (whole population, with risk factor, without risk factor) | from 22nd Dec 2023 to 30th Apr 2024 and from 22nd Dec 2024 to 30th Apr 2025
Number of subjects in both cohorts who were treated with antibiotics/antivirals during respiratory tract infections of the whole observation period (whole population, with risk factor, without risk factor) | from 22nd Dec 2023 to 30th Apr 2024 and from 22nd Dec 2024 to 30th Apr 2025
Number of subjects in both cohorts who were treated with antibiotics/antivirals during respiratory tract infections of the first observation period (whole population, with risk factor, without risk factor) | from 22nd Dec 2023 to 30th Apr 2024
Number of subjects in both cohorts who were treated with antibiotics/antivirals during respiratory tract infections of the second observation period (whole population, with risk factor, without risk factor) | from 22nd Dec 2024 to 30th Apr 2025
Description of severity of respiratory tract infections during the whole observation period in both cohorts (whole population, with risk factor, without risk factor) | from 22nd Dec 2023 to 30th Apr 2024 and from 22nd Dec 2024 to 30th Apr 2025

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Bonini, Professor, Principal Investigator — Institute of Translational Pharmacology, Italian National Research Council (IFT-CNR)
Locations (23):
- Italy (23):
  - Dr F Pugliese, Bari
  - Università degli Studi di Cagliari, Cagliari
  - Università degli studi di salerno, Fisciano
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Dr M D'Onofrio, Napoli
  - Azienda Ospedale Università Padova, Padua
  - Azienda Ospedale-Università Padova, Padua
  - Dr F Gatti, Parma
  - A.S.L. di Pescara - Abruzzo, Popoli
  - Dr F R Amorosi, Roma
  - Dr G Marrocco, Roma
  - Dr S Narzisi, Roma
  - Dr A Galli, Roma
  - Dr C Governale, Roma
  - Dr E Meco, Roma
  - Dr A M Pistuddi, Roma
  - Dr R Chini, Roma
  - Università Cattolica del Sacro Cuore, Roma
  - Dr G Biondi, Roma
  - Dr C Nicoletta, Salerno
  - Azienda Ospedaliera Mauriziano di Torino, Torino
  - ASST dei Sette Laghi, Varese
  - ASP Vibo Valentia, Vibo Valentia